CLINICAL TRIAL: NCT05279118
Title: Comparison of Efficacy of Ketogenic Diet and ACTH Therapy Among Children With West Syndrome: A Pilot Randomized Control Trial
Brief Title: Ketogenic Diet vs ACTH for the Treatment of Children With West Syndrome
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: All India Institute of Medical Sciences (Other)
Responsible Party: Principal Investigator, Sheffali Gulati, Professor, All India Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IECPG-19/27.1.2022,RT/24.2.22; No.3/2/June2022/PG-Thesis (Other Grant/Funding Number: ICMR)
Record Dates: First submitted 2022-03-03; First posted 2022-03-15 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Ketogenic Diet; West Syndrome; Infantile Spasm; ACTH
Keywords: Ketogenic diet; West Syndrome; Infantile Spasm; ACTH
MeSH Terms: conditions — Spasms, Infantile | interventions — Diet, Ketogenic; Diet Therapy; Adrenocorticotropic Hormone

STUDY DESIGN:
Intervention Model Description: pilot randomized RCT
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ketogenic diet arm (Experimental): Children who have consented to the study and have been randomised to ketogenic diet arm will get ketogenic diet under supervision while starting with rapid hiking of lipid to carbohydrate ratio and primary response will be assessed at 6 weeks. Ketogenic diet ratio will be hiked quickly upto a maximum of 4:!. The duration of ketogenic diet can be extended beyond the period of study based on response and parental choice. A minimum period of 6 weeks of diet therapy will be undertaken baring any undue adverse effects when the primary outcome will be assessed
  Interventions: Dietary Supplement: Ketogenic diet
- ACTH arm (Active Comparator): ACTH is the current standard therapy for children with west syndrome. Those who have been randomised to this arm will be started on high dose ACTH for 2 weeks followed by gradual tapering over remaining 4 weeks and primary response documented at 6 weeks of therapy. The high dose ACTh is 150U/m2 or 6U/kg dose administered IM daily for two weeks. After this the doses will be tapered gradually and ACTH will be stopped by 4 weeks for a total treatment duration of strictly 6 weeks.
  Interventions: Drug: ACTH

INTERVENTIONS:
Dietary Supplement: Ketogenic diet — Children who have consented to the study and have been randomised to ketogenic diet arm will get ketogenic diet under supervision while starting with rapid hiking of lipid to carbohydrate ratio and primary response will be assessed at 6 weeks. Ketogenic diet ratio will be hiked quickly upto a maximum of 4:!. The duration of ketogenic diet can be extended beyond the period of study based on response and parental choice. A minimum period of 6 weeks of diet therapy will be undertaken baring any undue adverse effects when the primary outcome will be assessed
  Other Names: Diet therapy
  Arms: Ketogenic diet arm
Drug: ACTH — ACTH is the current standard therapy for children with west syndrome. Those who have been randomised to this arm will be started on high dose ACTH for 2 weeks followed by gradual tapering over remaining 4 weeks and primary response documented at 6 weeks of therapy. The high dose ACTh is 150U/m2 or 6U/kg dose administered IM daily for two weeks. After this the doses will be tapered gradually and ACTH will be stopped by 4 weeks for a total treatment duration of strictly 6 weeks.
  Other Names: Hormonal therapy
  Arms: ACTH arm

SUMMARY:
Children with West syndrome are prone to refractory seizures with poor neurocognitive outcome overall. The current standard of care consists of treatment with ACTH, but the grade of evidence is not high and not much RCTs are available. Ketogenic diet is an effective and well tolerated treatment option in drug refractory epilepsy and also in refractory west syndrome. In view of minimal side effects, better cost parameters and ability to continue for a longer duration our study aiims to investigate the efficacy of ketogenic diet as a first line therapy in comparison to ACTH therapy. Children with west syndrome after satisfying the inclusion and exclusion criteria will be randomised into the two treatment arms and primary response will be noted at the end of 6 weeks of therapy in terms of mean percentage of spasm reduction.

DETAILED DESCRIPTION:
* Consecutive children with West Syndrome (clinical spasm with EEG correlate) will be screened in the study centre for eligibility, and after applying inclusion and exclusion criteria they will be worked up for etiology.
* History will be taken and clinical examination will be done and if either are suggestive of any underlying etiology specific investigations will be performed as indicated (Ex. Neurocutaneous markers in tuberous sclerosis).
* If there are no other etiological pointers available from history and examination or if there is any history suggestive of adverse perinatal events, MRI brain with epilepsy protocol will be done.
* If MRI is not suggestive of structural etiology they will be given a vitamin trial(pyridoxine 30mg/kg/day, pyridoxal phosphate- 20mg/kg/day, biotin 10mg/day and folinic acid 15mg/day) for a period of 10 days for response. Those who respond to Vitamin trial will be excluded from the study.
* Written informed consent will be taken from legal guardians who are willing to participate in the study. Their anti-epileptic drugs will be optimised. Inappropriate AEDs like phenytoin, phenobarbitone and carbamazepine will be discontinued and replaced with valproate/levetiracetam and clonazepam in adequate doses and will be made in tablet form.
* There will be an observation period of 2 weeks where the participants will be sensitised about proper counting of spasms and the mean no. of spasms per week of the 2nd week will form the baseline and they will be randomised into two groups as mentioned above during the same period with no further changes in AEDs till the duration of completion of primary objective. Those who require hiking/titrating of AEDs during the initial period of 6 weeks plus run in period of 2 weeks will be treated as deviates and excluded from the study.
* DASII will be administered by child psychologist and will be repeated at 3 months and at 6 months of followup wherever feasible.
* Appropriate screening for Tuberculosis as per unit protocol (Mantoux and CXR screening) will be done if going to the ACTH therapy arm.
* Workup for ketogenic diet will also be done ECG, RFT, LFT, CBC, Lipid profile, Urine calcium creatinine ratio and USG KUB for nephrocalcinosis if going to the KD arm

Group 1 ACTH arm:

* Children randomised into ACTH arm will be started on high dose regimen(45)(46) of 150U/m2 or 6U/kg of ACTH.
* This high dose will be continued for 2 weeks following which they will be slowly tapered over remaining 4 weeks, for a total treatment duration of 6 weeks.
* EEG will be done at 6 weeks and 3 months of therapy in case of clinical spasm cessation and wherever clinically indicated
* First followup will be at 6 weeks of treatment initiation, then at 8 weeks and from then on once a month for a minimum period of 3 months (+/- 7 days) upto 6 months(+/- 7 days) wherever feasible.
* Those who have had complete electroclinical spasm cessation will be continued of oral AEDs.
* Those who have <50% spasm reduction rate will be shifted to KD.
* Those who have >/=50% spasm reduction rate will be given trial of other oral AEDs as per protocol.
* The overall spasm reduction will be calculated from the mean number of spasms from the observation period week and the mean number of spasms from the 6th week of therapy. Adverse effects will be noted down in their seizure diary.
* For sustained electroclinical cessation those who had complete electroclinical response will be rechecked at the end of 3 months (+/- 7 days) upto 6 months(+/- 7 days) wherever feasible.
* Compliance rate, adverse events, >50% spasm reduction rate, clinical spasm cessation rate, complete electroclinical spasm cessation rate will also be calculated from patient seizure log and EEG correlate.
* RBS and BP monitoring to be done twice weekly

Group 2 KD arm:

* Children randomised into this arm will be admitted in ward and initiated on Ketogenic diet under supervision.
* KD will be initiated in a ratio of 2:1 and then hiked to 2.5:1 in the next day and subsequently to 3:on day 3. Urine ketones will be checked daily using ketone dipsticks.
* For better assurance of ketosis and tolerance the indigenous KD will be supplemented with readymade formula for the initial period of 4 weeks and then shifted to complete indigenous KD gradually over 1 week.
* If ketosis is not achieved by day 5 of starting KD, the ratio will be hiked to a maximum of 4:1 from day 6.
* Patient will be discharged as soon as the desired ratio of KD is achieved, and the parents are adequately motivated and confident. Telephonic contacts will be made in regular intervals to further ensure compliance at home.
* Those children who are unable to tolerate taking adequate ketogenic diet therapy requiring discontinuation of therapy, will be considered as deviates.
* The overall spasm reduction will be calculated from the mean number of spasms from the observation period week and the mean number of spasms from the 4th week of therapy.
* Failure of KD: Children with response rate if not >50% spasm reduction by 6 weeks or no electroclinical cessation of spasm by 3 months, will be considered to have failed KD and shifted to standard ACTH therapy as per protocol.
* KD will be continued if there is more than 50% spasm reduction.
* EEG will be done at 6 weeks and 3 months of therapy in case of clinical spasm cessation and wherever clinically indicated
* First followup will be at 6 weeks of treatment initiation,8weeks and then once monthly for a minimum period of 3 months and 6 months wherever feasible. For sustained electroclinical cessation those who had complete electroclinical response will be rechecked at the end of 3 months (+/- 7 days) upto 6 months(+/- 7 days) wherever feasible.
* Compliance rate, adverse events, >50% spasm reduction rate, clinical spasm cessation rate, complete electroclinical spasm cessation rate will also be calculated from patient seizure log and EEG correlate. .
* Formula based KD would be supplied to the patient free of cost. But the company will play no part in the study design, conduct, data collection or analysis

ELIGIBILITY:
Inclusion Criteria:

* Children, aged 6 month - 2 years with electroclinical diagnosis of west syndrome

Exclusion Criteria:

* Already on ACTH, prednisolone vigabatrin or KD therapy > 5days
* Tuberous sclerosis
* Vitamin trial responsiveness
* Known Pre-existing contraindications for KD (IEM, Porphyria etc.)
* Chronic systemic illness (Ex: Chronic kidney disease, congenital heart diseases etc)

Ages: 6 Months to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2022-04-18 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2024-07-28 (Estimated)

PRIMARY OUTCOMES:
Mean percentage reduction of spam (Baseline mean weekly spasm rate - mean weekly spasm rate on 6th week of therapy/Baseline mean weekly spasm rate * 100) is compared in both arms | From baseline to 6 weeks of therapy
  Mean percentage reduction of spam (Baseline mean weekly spasm rate - mean weekly spasm rate on 6th week of therapy/Baseline mean weekly spasm rate * 100) is compared in both arms

SECONDARY OUTCOMES:
To compare complete spasm cessation rate in KD arm vs ACTH arm | Percentage of children with clinical spasm cessation at 6 weeks of therapy
  Percentage of children with clinical spasm cessation at 6 weeks of therapy
To compare >50% spasm reduction rate in KD arm vs ACTH arm | Percentage of children with >50% spasm reduction at the end of 6 weeks and 3months of therapy (wherever feasible at 6 months)
  Percentage of children with >50% spasm reduction at the end of 6 weeks and 3months of therapy (wherever feasible at 6 months)
To compare electroclinical spasm To compare electroclinical spasm cessation rate in KD arm vs ACTH arm at 6 weeks | Percentage of children with clinical spasm cessation at 6 weeks of therapy
  Percentage of children with clinical spasm cessation at 6 weeks of therapy
To compare sustained electroclinical cessation rate in KD arm vs ACTH arm at 3 months | Percentage of children with primary electroclinical spasm cessation who sustain the remission at 3months of therapy(wherever feasible at 6 months)
  Percentage of children with primary electroclinical spasm cessation who sustain the remission at 3months of therapy(wherever feasible at 6 months)
To compare the compliance rate in KD arm vs ACTH arm at 6 weeks | Percentage of children with compliance of greater than >80% of doses of ACTH in the 6 weeks of therapy compared with percentage of children with score of >80% in KD compliance questionnaire (score of >/=18 out of 25)
  Percentage of children with compliance of greater than >80% of doses of ACTH in the 6 weeks of therapy compared with percentage of children with score of >80% in KD compliance questionnaire (score of >/=18 out of 25)
To compare the adverse effect profile in KD arm vs ACTH arm at 6 weeks and 3 months | Description of adverse effects in each groups with proportion of CTCAE grade 3 and above in each groups at 3months of therapy (wherever feasible at 6 months)
  Description of adverse effects in each groups with proportion of CTCAE grade 3 and above in each groups at 3months of therapy (wherever feasible at 6 months)
To compare neurodevelopmental outcome in KD arm vs ACTH arm using DASII at 3 months | Percentage improvement in Motor and Mental developmental quotients of children in both groups at 3 months of therapy (wherever feasible at 6 months)
  Percentage improvement in Motor and Mental developmental quotients of children in both groups at 3 months of therapy (wherever feasible at 6 months)

CONTACTS AND LOCATIONS:
Overall Officials: Sheffali Gulati, Principal Investigator — All India Institute of Medical Sciences
Locations (2):
- India (2):
  - All India Institute of Medical Sciences, New Delhi, National Capital Territory of Delhi
  - AIIMS, New Delhi

IPD SHARING:
Plan to Share IPD: No